CLINICAL TRIAL: NCT03135509
Title: A Phase 1, Open-label, Single-center Study to Assess the Relative Bioavailability of a New CC-220 Capsule Formulation, Compared to a Reference CC-220 Capsule Formulation, in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability of a New CC-220 Capsule Formulation, Compared to a Reference CC-220 Capsule Formulation, in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-CP-005; U1111-1195-6929 (Registry Identifier: WHO)
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy Subjects; CC-220 Capsules; Relative Bioavailability; Phase 1
MeSH Terms: interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Reference)- CC-220 gelatin capsules (Experimental): A single dose of 0.6 mg CC-220, administered as two 0.3-mg formulated CC-220 gelatin capsules.
  Interventions: Drug: CC-220
- Treatment B (Test)- CC-220 HPMC capsule (Experimental): A single dose of 0.6 mg CC-220, administered as one 0.6-mg formulated CC-220 hydroxypropyl methylcellulose (HPMC) capsule.
  Interventions: Drug: CC-220

INTERVENTIONS:
Drug: CC-220 — CC-220 gelatin capsules

SUMMARY:
This is an open-label, randomized, 2-period, 2-way crossover study to assess the relative bioavailability of a new CC-220 capsule formulation, compared to a reference CC-220 capsule formulation, after administration of single oral doses in healthy adult subjects under fasted conditions.

Approximately 16 subjects will be assigned randomly to 1 of 2 treatment sequences. The sequences will dictate the order in which each subject receives the following treatments:

* Treatment A (Reference): A single dose of 0.6 mg CC-220, administered as two 0.3-mg formulated CC-220 gelatin capsules.
* Treatment B (Test): A single dose of 0.6 mg CC-220, administered as one 0.6-mg formulated CC-220 Hydroxypropyl methylcellulose (HPMC) capsule.

DETAILED DESCRIPTION:
The study will consist of 2 study periods. Each subject will participate in a screening phase, a baseline phase in each study period, a treatment phase in each study period, and a follow up telephone call. Subjects will be screened for eligibility. Eligible subjects will return to the study center on Day -1 of Period 1, and will remain domiciled at the study center from Day -1 of Period 1 to Day 4 of Period 2.

On Day 1 of Period 1, eligible subjects will be randomized to 1 of 2 sequences. On Day 1 of each study period, each subject will receive 1 of 2 treatments according to the sequence in which he or she is randomized.

Blood samples will be collected at prespecified times for PK, PD, and clinical laboratory safety tests. Urine samples will be collected at prespecified times for clinical laboratory safety tests.

Safety will be monitored throughout the study. Safety evaluations will include AE reporting, review of concomitant medications and procedures, physical examinations (PEs), 12-lead ECGs, vital sign measurements, and clinical laboratory safety tests. Subjects will be discharged from the study center on Day 4 of Period 2 upon completion of scheduled study-related procedures and satisfactory safety review. Each subject will receive a follow-up telephone call within 5 to 7 days following discharge from the study center.

The study will be conducted in compliance with the International Council on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 and ≤ 65 years of age at the time of signing the Informed Consent Form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health, as determined by the Investigator based on a Physical examination (PE) at screening.
5. Subject agrees to abide by the requirements and restrictions outlined in the CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
6. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).
7. Male subjects must:

   a. Practice true abstinence1 (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or female of childbearing potential (FCBP)2 while participating in the study, during dose interruptions, and for at least 90 days after the last dose of investigational product (IP), even if he has undergone a successful vasectomy.
8. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator. Platelet count, absolute neutrophil count, and absolute lymphocyte count must be above the lower limit of normal at screening.
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    1. If male, subject has a QTcF value ≤ 430 msec at screening.
    2. If female, subject has a QTcF value ≤ 450 msec at screening.

Exclusion Criteria:

Inclusion Criteria: DO NOT USE ACROYNMS

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 and ≤ 65 years of age at the time of signing the Informed Consent Form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health, as determined by the Investigator based on a Physical examination (PE) at screening.
5. Subject agrees to abide by the requirements and restrictions outlined in the CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
6. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle- stimulating hormone [FSH] level of > 40 IU/L at screening).
7. Male subjects must:

   a. Practice true abstinence1 (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or female of childbearing potential (FCBP)2 while participating in the study, during dose interruptions, and for at least 90 days after the last dose of investigational product (IP), even if he has undergone a successful vasectomy.
8. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator. Platelet count, absolute neutrophil count, and absolute lymphocyte count must be above the lower limit of normal at screening.
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    1. If male, subject has a QTcF value ≤ 430 msec at screening.
    2. If female, subject has a QTcF value ≤ 450 msec at screening.

Exclusion Criteria: DO NOT USE ACROYNMS

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is a female of childbearing potential, pregnant, or breastfeeding.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
6. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 14 days or 5 half-lives of that medication, whichever is longer, prior to the first dose administration.
7. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 7 days prior to the first dose administration.
8. Subject has used Cytochrome P450 (CYP)3A inducers and/or inhibitors (including St. John's wort) within 30 days prior to the first dose administration..
9. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable.
10. Subject donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
11. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive drug test reflecting consumption of illicit drugs.
12. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years before the first dose administration, or positive alcohol test.
13. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
14. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
15. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to administration of the first dose of IP or is planning to receive immunization with a live or live attenuated vaccine for 2 months after administration of the last dose of IP.
16. Subject is part of the clinical staff personnel or a family member of the clinical site staff.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
PK - Cmax | Up to approximately 1 month
  Observed maximum plasma concentration
PK - AUC0-t | Up to approximately 1 month
  Area under the concentration-time curve calculated from time zero to the last measured time point

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 1 month
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, MD, Study Director — Celgene Corporation
Locations (1):
- Quintiles Phase One Services, LLC, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No